CLINICAL TRIAL: NCT06933381
Title: Topical Vapocoolant to Reduce Pain With Nexplanon Insertion: A Randomized Controlled Trial
Brief Title: Vapocoolant Spray to Reduce Pain With Nexplanon Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: Lakshmi Devi and Devraj Sharma Endowment (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RA-2025-007
Record Dates: First submitted 2025-03-31; First posted 2025-04-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Reducing Pain With Nexplanon Implant Insertion
Keywords: Vapocoolant spray; Pain with Nexplanon insertion; Contraceptive implant insertion; Vapocoolant

STUDY DESIGN:
Who Masked: Participant
Masking Description: Research coordinators collecting pain scales from patients will also be blinded to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vapocoolant Spray (Experimental): This is the study arm. Participants in this arm of the study will receive Pain Ease vapocoolant spray during their Nexplanon implant insertion in the arm. They will receive the spray on their arm right before lidocaine injection is administered for Nexplanon insertion procedure. Pain Ease vapocoolant spray is FDA approved for use on skin prior to common needle-stick procedures like intravenous (IV) starts and vaccines. The investigators will use the spray in a similar fashion, to help with the pain of lidocaine injection during Nexplanon insertion procedures. Physicians will do the Nexplanon procedure before any other procedures if patient has multiple procedures scheduled the same day.
  Interventions: Device: Vapocoolant spray
- Nature's Tears (Placebo Comparator): This is the placebo. This group will receive Nature's Tears, which is a saline spray that does not offer analgesic effects.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Vapocoolant spray — Pain Ease will be used per manufacturer instruction, applying the spray for 5 seconds or until the skin turns white, whichever occurs first.
  Other Names: Pain Ease
  Arms: Vapocoolant Spray
Other: Placebo — Nature's Tears will be applied to the arm as a placebo spray
  Other Names: Nature's Tears
  Arms: Nature's Tears

SUMMARY:
The purpose of this study is to assess if Pain Ease vapocoolant spray decreases pain associated with lidocaine injection during Nexplanon insertion procedures.

DETAILED DESCRIPTION:
This study will be for patients in the office having a Nexplanon (etonogestrel implant) insertion. The doctor in clinic will evaluate if a patient meets eligibility criteria for this study. If the patient meets eligibility criteria, the doctor will inform the patient of the study and the potential risks. If patients elect to participate, a research coordinator will obtain written informed consent. The patient will be randomized (patient is blinded) to receive either Pain Ease vapocoolant spray or placebo (normal saline) spray. They will receive the spray just before lidocaine injection during the Nexplanon insertion procedure. The purpose of the study is to see if Pain Ease vapocoolant spray reduces patient pain during lidocaine injection for Nexplanon insertion.

ELIGIBILITY:
Inclusion Criteria:

* At least 14 years or older
* Undergoing an etonogestrel implant insertion in the arm in POB1 Suite 1004 or POB2 Suite 402
* English speaking
* Able and willing to sign the informed consent form and agree to terms of the study

Exclusion Criteria:

* Required or requested narcotics, anxiolytics, IV sedation, or general anesthesia for the procedure
* Known previous exposure to vapocoolant spray
* Nexplanon removal and reinsertion same day during visit in the same arm
* Contraindications to vapocoolant spray components (ethyl chloride and 1,1,1,3,3-pentafluoropropane/1,1,1,2-tetrafluroethane)
* Unable to provide written, informed consent in English

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain with lidocaine injection | Immediately after lidocaine injection
  The investigators will ask patients to rate their pain with lidocaine injection that precedes Nexplanon insertion using a visual analog scale (VAS). The visual analog scale is a 100 mm line, with values 0 to 100. 0 is marked as no pain and 100 is marked as worst pain.

SECONDARY OUTCOMES:
Patient satisfaction | Immediately after procedure
  Patients will be asked about their satisfaction with pain control for the procedure and satisfaction for the procedure overall using a survey with 5 options, including very unsatisfied, unsatisfied, neutral, satisfied, and very satisfied.
Pain Reduction with Remainder of Procedure | Immediately after the procedure
  Participants will be asked to rate their pain using a visual analog scale (VAS) in regard to pain when the implant was inserted. The visual analog scale is a 100 mm line, with values 0 to 100. 0 is marked as no pain and 100 is marked as worst pain.They will also be asked about their pain for the procedure overall using a Likert scale from 0 (no pain) to 10 (severe pain).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Queens Medical Center POB 2 Suite 402, Honolulu, Hawaii
  - Queens Medical Center POB1 Clinic 1004, Honolulu, Hawaii
  - Women's Center Queen's North Hawai'i Community Hospital Suite #124 and #120, Waimea, Hawaii

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Mace SE. Prospective, randomized, double-blind controlled trial comparing vapocoolant spray vs placebo spray in adults undergoing venipuncture. Am J Emerg Med. 2016 May;34(5):798-804. doi: 10.1016/j.ajem.2016.01.002. Epub 2016 Jan 7. PMID 26979261
- [Background] Unal N, Tosun B, Aslan O, Tunay S. Effects of Vapocoolant Spray Prior to SC LMWH Injection: An Experimental Study. Clin Nurs Res. 2021 Feb;30(2):127-134. doi: 10.1177/1054773818825486. Epub 2019 Jan 30. PMID 30698458
- [Background] Zhu Y, Peng X, Wang S, Chen W, Liu C, Guo B, Zhao L, Gao Y, Wang K, Lou F. Vapocoolant spray versus placebo spray/no treatment for reducing pain from intravenous cannulation: A meta-analysis of randomized controlled trials. Am J Emerg Med. 2018 Nov;36(11):2085-2092. doi: 10.1016/j.ajem.2018.03.068. Epub 2018 Mar 27. PMID 30253890
- [Background] Collado-Mesa F, Net JM, Arheart K, Klevos GA, Yepes MM. Application of a topical vapocoolant spray decreases pain at the site of initial intradermal anaesthetic injection during ultrasound-guided breast needle biopsy. Clin Radiol. 2015 Sep;70(9):938-42. doi: 10.1016/j.crad.2015.04.013. Epub 2015 Jul 7. PMID 26162573
- [Background] Wilson GA, Jeter JW, Dabbs WS, Stevens AB, Heidel RE, Chamberlin SM. Comparison of traditional anesthesia method and jet injector anesthesia method (MadaJet XL(R)) for Nexplanon(R) insertion and removal. Contracept Reprod Med. 2020 Feb 24;5:1. doi: 10.1186/s40834-020-00104-x. eCollection 2020. PMID 32123573
- [Background] Bentsianov SD, Brandi K, Chen P, Shimoni N. A Pilot Study to Understand the Adolescent Pain Experience During Contraceptive Implant Insertion. J Pediatr Adolesc Gynecol. 2021 Aug;34(4):522-524. doi: 10.1016/j.jpag.2021.01.013. Epub 2021 Jan 27. PMID 33515699
- See also: Gebauer's Pain Ease — https://www.gebauer.com/painease?utm_term=pain%20ease&utm_campaign=Pain+Ease+-+Branded&utm_source=adwords&utm_medium=ppc&hsa_acc=7587893839&hsa_cam=1585937464&hsa_grp=58836587414&hsa_ad=647795903980&hsa_src=g&hsa_tgt=kwd-306943226566&hsa_kw=pain%20ease&hsa_mt=e&hsa_net=adwords&hsa_ver=3&gad_source=1&gclid=Cj0KCQiAlbW-BhCMARIsADnwaspKAF4-pot2OT1xRBDi-6mPr1B4ixzm5SPWAy6mhKPzWFaisRe1p90aAqvVEALw_wcB